CLINICAL TRIAL: NCT06778005
Title: Investigation of the Relationship of Ultrasonographic Measurements of Lower Extremity Nerves With Gait and Balance Performance in Type 2 Diabetes Patients With Peripheral Polyneuropathy
Brief Title: Investigation of Ultrasonographic Measurements of Lower Extremity Nerves in Type 2 Diabetes Patients With Peripheral Polyneuropathy
Status: Recruiting | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 14/2
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-05

CONDITIONS: Diabetes; Diabetic Polyneuropathy
Keywords: polyneuropathy; Ultrasound; diabetes; balance; gait
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies; Polyneuropathies | interventions — Ultrasonography; Walk Test; Physical Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Healthy volunteers): Healthy volunteers without diabetes diagnosis will be included in group 1. (n=17)
  Interventions: Diagnostic Test: Ultrasonography; Diagnostic Test: Biodex Balance System; Diagnostic Test: Douleur Neuropathique 4 (DN4) Pain Scale; Diagnostic Test: Numeric Rating Scale; Diagnostic Test: Toronto Clinical Neuropathy Score; Diagnostic Test: Six-Minute Walk Test; Diagnostic Test: SF-12 Quality of Life Scale; Combination Product: International Physical Activity Questionnaire-Short Form (IPAQ); Diagnostic Test: Tuning Fork Vibration Sense; Diagnostic Test: Timed Up and Go Test; Diagnostic Test: Physical Examination
- Group 2 ( Patients with diabetic polyneuropathy): Patients with diabetic polyneuropathy will be included in group 2. (n=69)
  Interventions: Diagnostic Test: Ultrasonography; Diagnostic Test: Biodex Balance System; Diagnostic Test: Douleur Neuropathique 4 (DN4) Pain Scale; Diagnostic Test: Numeric Rating Scale; Diagnostic Test: Toronto Clinical Neuropathy Score; Diagnostic Test: Six-Minute Walk Test; Diagnostic Test: SF-12 Quality of Life Scale; Combination Product: International Physical Activity Questionnaire-Short Form (IPAQ); Diagnostic Test: Tuning Fork Vibration Sense; Diagnostic Test: Timed Up and Go Test; Diagnostic Test: Physical Examination

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Measurements will be performed using a 7-12 MHz Sonosite M-Turbo device (Fujifilm, USA) with a linear probe by an operator trained in peripheral nervous system ultrasonography. Cross-sectional area (CSA) and echogenicity measurements of the bilateral tibial, common peroneal, and sural nerves will be conducted using the ultrasound device. Tibial nerve assessment will be performed 3 cm proximal to the level of the medial malleolus. Common peroneal nerve assessment will be performed by identifying the nerve at the fibular head and tracking it proximally to image it at the level of the popliteal fossa. Sural nerve assessment will be conducted 10 cm proximal to the upper level of the lateral malleolus. All nerve measurements will be conducted twice in the transverse plane, and the obtained images will be recorded and uploaded into the ImageJ programming system.
Diagnostic Test: Biodex Balance System — The Biodex is a computer-assisted device with a movement system capable of providing surface inclinations ranging from 360 degrees to 20 degrees. It allows movement in anterior/posterior and mediolateral planes. The device has 12 levels of difficulty, where level 12 represents the highest stability and level 1 represents the lowest stability. It can be used for balance training with different therapy protocols and includes standardized programming systems for evaluating both static and dynamic balance. It provides numerical data for key parameters such as balance, fall risk, and proprioception. In this study, patients will be assessed using the fall risk test and postural stability evaluation test protocols on the Biodex balance system. All participants will be trained and familiarized with the system before the test.
  Postural Stability Test: The difficulty level will be set to 8. Fall Risk Test: The difficulty level will progressively decrease from 6 to 2.
Diagnostic Test: Douleur Neuropathique 4 (DN4) Pain Scale — The Douleur Neuropathique 4 (DN4) pain scale score will be used to screen for diabetic peripheral neuropathic pain. The DN4 scale consists of 10 questions, 7 of which inquire about symptoms, and 3 that assess the patient's clinical examination for neuropathy. The symptoms assessed include a burning sensation, pain from cold, electric shock sensations, tingling, pins and needles, numbness, and itching. The sensory exams assess touch hypoesthesia, pin-prick hypoesthesia, and brush allodynia. Each "yes" response to a question receives 1 point. To calculate the total score, points obtained from the symptom inquiry and clinical examination are added together. The maximum total score is 10, and a score of 4 or higher is considered indicative of neuropathic pain
Diagnostic Test: Numeric Rating Scale — The numeric pain scale will be used to assess the intensity of neuropathic pain. The patient is asked to provide a value between 0 and 10 to indicate the intensity of their pain. Higher scores are associated with an increase in pain severity.
Diagnostic Test: Toronto Clinical Neuropathy Score — The Toronto Clinical Neuropathy Score (TCNS) will be used to assess the severity of Diabetic Peripheral Polyneuropathy (DPPN). The Turkish version of the Toronto clinical scoring system is a reliable and valid tool for assessing polyneuropathy in Turkish-speaking patients. The TCNS is preferred in clinical studies because of its ease of use, patient acceptability, ability to classify the severity of DPPN, and its representation of clinical changes related to the progression of DPPN. The scale consists of three sections: symptom scores, sensory test scores, and reflex scores.The first section includes scoring symptoms in the upper and lower extremities .The second section includes scoring the bilateral Achilles and patellar reflexes. The third section involves scoring the sensation in the toe. The total score ranges from a minimum of 0 (no neuropathy) to a maximum of 19 points.
Diagnostic Test: Six-Minute Walk Test — Six-Minute Walk Test (6MWT) is a commonly used test to assess functional capacity. The test area should be a corridor with a minimum length of 30 meters, flat, and firm surface. The corridor should be marked every 3 meters. Turnaround points are indicated with objects such as orange traffic cones. A line is drawn for the start and end of the test. Recommended materials for the test include a stopwatch, a device to count laps, cones to mark turning points, a chair placed within easy reach, oxygen support (to be given if necessary), and a blood pressure cuff. The patient should wear comfortable clothing and shoes suitable for walking. They can use any walking aids such as crutches or a walker. Medications or treatments should be taken as usual. The patient should have had a light meal before the test and should not have engaged in heavy physical activity within the 2 hours preceding the test. There should be no warm-up period before the test.
Diagnostic Test: SF-12 Quality of Life Scale — The SF-12 Quality of Life Scale will be calculated using an online calculator tool, providing two types of scores: physical and mental scores.
Combination Product: International Physical Activity Questionnaire-Short Form (IPAQ) — The IPAQ scale was developed to address the general health problem of insufficient physical activity, which necessitates large population studies and allows for cross-country comparisons. Validity studies conducted across multiple countries have proven that this questionnaire is valid and reliable. This survey assesses individuals based on the types of physical activities they perform in their daily lives. The questions asked pertain to the time spent physically active over the past 7 days.
Diagnostic Test: Tuning Fork Vibration Sense — Vibration sense will be assessed using a traditional 128 Hz tuning fork. When the stem of a 128 Hz tuning fork is placed on the dorsal aspect of the interphalangeal joint of the hallux, a healthy person can feel the vibration as long as it continues (15-20 seconds). In conditions leading to peripheral nerve damage (such as polyneuropathy), vibration sense is impaired. The examiner holds the proximal end of the tuning fork with one hand, while the distal end is struck strongly against the palm of the examiner's other hand. The examiner should try to strike the tuning fork with consistent force for each assessment. After striking, the tuning fork is placed just proximal to the nail bed, on the dorsal aspect of the distal phalanx of the hallux.Before applying the tuning fork, the participant is instructed to verbally respond with "yes" if they can initially feel the vibration, and they should also indicate "now" when they stop feeling the vibration.
Diagnostic Test: Timed Up and Go Test — The Timed Up and Go (TUG) test is designed to measure dynamic balance based on the time it takes for patients to stand up and walk, providing quantitative results. The patient starts the test by sitting on a standardized chair (46 cm high). During the test, the patient is instructed to stand up from the chair, walk 3 meters away, turn around, and then return to sit back down on the chair. The duration of this process is measured. Lower values indicate better stability. A cutoff value of 13.5 seconds has been used to identify high fall risk in the TUG test.
Diagnostic Test: Physical Examination — Manual Muscle Test: Muscle strength is evaluated using the MRC (Medical Research Council) muscle strength scale.
  Reflexes:Patellar reflex: The reflex hammer is struck on the patella, and extension of the leg is observed. Achilles reflex: With one hand, the patient's foot is lightly dorsiflexed, and the Achilles tendon is struck; plantar flexion is observed in the ankle.

SUMMARY:
The aim of this study is to quantitatively evaluate ultrasonographic measurements of the lower extremity nerves in patients diagnosed with diabetic polyneuropathy and to investigate the relationship with gait, static and dynamic balance performance.

In this study, we aimed to investigate the effect of ultrasonographic findings of lower extremity nerves on quality of daily life, physical activity, gait and balance in patients with diabetic peripheral polyneuropathy.

DETAILED DESCRIPTION:
Diabetes is a chronic metabolic disorder characterized by hyperglycemia and the body's inability to adequately utilize carbohydrates, fats, and proteins due to a reduction in insulin secretion or insulin action. It requires continuous medical care.

One of the most common complications associated with diabetes is diabetic neuropathy, which affects the autonomic, motor, and sensory nerves of the peripheral nervous system. The most frequent form of diabetic neuropathy is peripheral sensorimotor polyneuropathy. Clinical and electrophysiological findings typically begin in the distal lower extremities.

While nerve conduction studies remain the gold standard for diagnosing diabetic neuropathy, they are time-consuming, require a separate patient visit, and are too costly to recommend for routine screening. Various methods can be employed to assess the morphological changes in nerves associated with diabetic peripheral neuropathy. With advancing technology in recent years, ultrasonography (US) has emerged as an affordable, reproducible, and more comfortable technique. It can be utilized as an effective method to evaluate structural changes in nerves. Diabetic neuropathy is a significant contributor to the severe morbidity, increased mortality, and reduced quality of life in diabetic patients. Therefore, the early detection of nerve dysfunction through ultrasonography is essential for providing appropriate care to patients with diabetic neuropathy.

The study will be conducted as a cross-sectional and single-center research involving patients with peripheral polyneuropathy secondary to type 2 diabetes and healthy volunteers who present to the Physical Medicine and Rehabilitation Clinic at the Health Sciences University Sultan 2nd Abdülhamid Han Training and Research Hospital.

As part of the study, demographic data collected from participants will include age, gender, height, weight, body mass index, smoking and alcohol usage, marital status, occupation, educational level, fasting blood glucose, HbA1c levels, vitamin B12, ALT, AST, creatinine levels, duration of diabetes, duration of diabetic peripheral polyneuropathy (DPP) complaints, current antidiabetic medications, presence of comorbidities, and neuropathic pain treatment and duration. Patients will be evaluated once, and the assessment will include ultrasonography, the Biodex balance system, the Douleur Neuropathique 4 (DN4) pain scale, numeric pain scale, Toronto Clinical Neuropathy Score, diapason vibration sensitivity test, 6-minute walk test, SF-12 quality of life scale, International Physical Activity Questionnaire-Short Form, Timed Up and Go Test (TUG), and motor and sensory examination.

The sample size for the study was calculated using G-Power version 3.1, based on ultrasonographic measurement data from a similar study conducted by Breiner et al. in 2016. The calculated sample size includes Group 1: 17 healthy participants of similar age and gender, and Group 2: 69 participants diagnosed with peripheral polyneuropathy and type 2 diabetes, amounting to a total of 86 participants. The study is planned to be conducted between December 2024 and May 2025.

ELIGIBILITY:
Inclusion Criteria (Group 1):

* Being between the ages of 18-65
* Being literate
* Signed a voluntary consent form agreeing to participate in the study

Inclusion Criteria (Group 2):

* Diagnosed with Type 2 Diabetes based on at least one of the following diagnostic criteria: fasting plasma glucose ≥ 126 mg/dl, 2-hour plasma glucose ≥ 200 mg/dl in an oral glucose tolerance test, HbA1c ≥ 6.5%, or diabetes symptoms (excessive thirst, eating, urination, and weight loss) + random plasma glucose ≥ 200 mg/dl. (14)
* Diagnosed with diabetic peripheral polyneuropathy through EMG evaluation in addition to Type 2 Diabetes.
* Being between the ages of 18-65
* Being literate
* Signed a voluntary consent form agreeing to participate in the study.

Exclusion Criteria:

* Individuals under 18 years old and over 65 years old
* Diagnosed with Type 1 diabetes
* Use of medications that can cause polyneuropathy
* Other causes of neuropathic pain (lumbar radiculopathy, spinal stenosis, -hereditary, inflammatory, entrapment neuropathies)
* Undergoing lower extremity surgery (spine/hip/knee/foot) in the last 6 months
* Having peripheral artery disease
* B12 vitamin deficiency
* Active foot ulcer
* History of lower extremity amputation
* Severe cardiopulmonary insufficiency (stage 3-4)
* History of myocardial infarction within the last 1 month
* History of unstable angina
* Active systemic inflammatory diseases and active malignancy
* Presence of vestibular disorders
* Presence of cognitive impairment
* Osteoarthritis in the lower extremity
* Pregnancy
* Body Mass Index (BMI) of 30 or higher

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic polyneuropathy and healthy volunteers aged between 18-65 years old will be evaluated visiting our physical medicine and rehabilitation outpatient clinic between December 2024 and May 2025.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasonography | 6 months
  Measurements will be performed using a 7-12 MHz Sonosite M-Turbo device (Fujifilm, USA) with a linear probe by an operator trained in peripheral nervous system ultrasonography. Cross-sectional area (CSA) and echogenicity measurements of the bilateral tibial, common peroneal, and sural nerves will be conducted using the ultrasound device. Tibial nerve assessment will be performed 3 cm proximal to the level of the medial malleolus. Common peroneal nerve assessment will be performed by identifying the nerve at the fibular head and tracking it proximally to image it at the level of the popliteal fossa. Sural nerve assessment will be conducted 10 cm proximal to the upper level of the lateral malleolus. All nerve measurements will be conducted twice in the transverse plane, and the obtained images will be recorded and uploaded into the ImageJ programming system.

SECONDARY OUTCOMES:
Biodex Balance System | 6 months
  The Biodex is a computer-assisted device with a movement system capable of providing surface inclinations ranging from 360 degrees to 20 degrees. It allows movement in anterior/posterior and mediolateral planes. The device has 12 levels of difficulty, where level 12 represents the highest stability and level 1 represents the lowest stability. It can be used for balance training with different therapy protocols and includes standardized programming systems for evaluating both static and dynamic balance. It provides numerical data for key parameters such as balance, fall risk, and proprioception. In this study, patients will be assessed using the fall risk test and postural stability evaluation test protocols on the Biodex balance system. All participants will be trained and familiarized with the system before the test. Postural Stability Test: The difficulty level will be set to 8. Fall Risk Test: The difficulty level will progressively decrease from 6 to 2.
Douleur Neuropathique 4 (DN4) Pain Scale | 6 months
  The Douleur Neuropathique 4 (DN4) pain scale score will be used to screen for diabetic peripheral neuropathic pain. The DN4 scale consists of 10 questions, 7 of which inquire about symptoms, and 3 that assess the patient's clinical examination for neuropathy. The symptoms assessed include a burning sensation, pain from cold, electric shock sensations, tingling, pins and needles, numbness, and itching. The sensory exams assess touch hypoesthesia, pin-prick hypoesthesia, and brush allodynia. Each "yes" response to a question receives 1 point. To calculate the total score, points obtained from the symptom inquiry and clinical examination are added together. The maximum total score is 10, and a score of 4 or higher is considered indicative of neuropathic pain
Numeric Rating Scale | 6 months
  The numeric pain scale will be used to assess the intensity of neuropathic pain. The patient is asked to provide a value between 0 and 10 to indicate the intensity of their pain. Higher scores are associated with an increase in pain severity.
Toronto Clinical Neuropathy Score | 6 months
  The Toronto Clinical Neuropathy Score (TCNS) will be used to assess the severity of Diabetic Peripheral Polyneuropathy (DPPN). The Turkish version of the Toronto clinical scoring system is a reliable and valid tool for assessing polyneuropathy in Turkish-speaking patients. The TCNS is preferred in clinical studies because of its ease of use, patient acceptability, ability to classify the severity of DPPN, and its representation of clinical changes related to the progression of DPPN. The scale consists of three sections: symptom scores, sensory test scores, and reflex scores.The first section includes scoring symptoms in the upper and lower extremities .The second section includes scoring the bilateral Achilles and patellar reflexes. The third section involves scoring the sensation in the toe. The total score ranges from a minimum of 0 (no neuropathy) to a maximum of 19 points.
Six-Minute Walk Test | 6 months
  Six-Minute Walk Test (6MWT) is a commonly used test to assess functional capacity. The test area should be a corridor with a minimum length of 30 meters, flat, and firm surface. The corridor should be marked every 3 meters. Turnaround points are indicated with objects such as orange traffic cones. A line is drawn for the start and end of the test. Recommended materials for the test include a stopwatch, a device to count laps, cones to mark turning points, a chair placed within easy reach, oxygen support (to be given if necessary), and a blood pressure cuff. The patient should wear comfortable clothing and shoes suitable for walking. They can use any walking aids such as crutches or a walker. Medications or treatments should be taken as usual. The patient should have had a light meal before the test and should not have engaged in heavy physical activity within the 2 hours preceding the test. There should be no warm-up period before the test.
SF-12 Quality of Life Scale | 6 months
  The SF-12 Quality of Life Scale will be calculated using an online calculator tool, providing two types of scores: physical and mental scores.
International Physical Activity Questionnaire-Short Form (IPAQ) | 6 months
  The IPAQ scale was developed to address the general health problem of insufficient physical activity, which necessitates large population studies and allows for cross-country comparisons. Validity studies conducted across multiple countries have proven that this questionnaire is valid and reliable. This survey assesses individuals based on the types of physical activities they perform in their daily lives. The questions asked pertain to the time spent physically active over the past 7 days.
Tuning Fork Vibration Sense | 6 months
  Vibration sense will be assessed using a traditional 128 Hz tuning fork. When the stem of a 128 Hz tuning fork is placed on the dorsal aspect of the interphalangeal joint of the hallux, a healthy person can feel the vibration as long as it continues (15-20 seconds). In conditions leading to peripheral nerve damage (such as polyneuropathy), vibration sense is impaired. The examiner holds the proximal end of the tuning fork with one hand, while the distal end is struck strongly against the palm of the examiner's other hand. The examiner should try to strike the tuning fork with consistent force for each assessment. After striking, the tuning fork is placed just proximal to the nail bed, on the dorsal aspect of the distal phalanx of the hallux.Before applying the tuning fork, the participant is instructed to verbally respond with "yes" if they can initially feel the vibration, and they should also indicate "now" when they stop feeling the vibration.
Timed Up and Go Test | 6 months
  The Timed Up and Go (TUG) test is designed to measure dynamic balance based on the time it takes for patients to stand up and walk, providing quantitative results. The patient starts the test by sitting on a standardized chair (46 cm high). During the test, the patient is instructed to stand up from the chair, walk 3 meters away, turn around, and then return to sit back down on the chair. The duration of this process is measured. Lower values indicate better stability. A cutoff value of 13.5 seconds has been used to identify high fall risk in the TUG test.
Physical Examination | 6 months
  Manual Muscle Test: Muscle strength is evaluated using the MRC (Medical Research Council) muscle strength scale. Reflexes:Patellar reflex: The reflex hammer is struck on the patella, and extension of the leg is observed. Achilles reflex: With one hand, the patient's foot is lightly dorsiflexed, and the Achilles tendon is struck; plantar flexion is observed in the ankle.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Ass. Prof., Study Director — Sultan 2. Abdulhamid Han Training and Research Hospital; Feyza Nur Yücel, Specialist, Study Director — Sultan 2. Abdulhamid Han Training and Research Hospital; Semiha Özgüç, M.D., Principal Investigator — Sultan 2. Abdulhamid Han Training and Research Hospital
Locations (1):
- Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bril V, Tomioka S, Buchanan RA, Perkins BA; mTCNS Study Group. Reliability and validity of the modified Toronto Clinical Neuropathy Score in diabetic sensorimotor polyneuropathy. Diabet Med. 2009 Mar;26(3):240-6. doi: 10.1111/j.1464-5491.2009.02667.x. PMID 19317818
- [Result] Arnold BL, Schmitz RJ. Examination of balance measures produced by the biodex stability system. J Athl Train. 1998 Oct;33(4):323-7. PMID 16558529
- [Result] Arumugam T, Razali SN, Vethakkan SR, Rozalli FI, Shahrizaila N. Relationship between ultrasonographic nerve morphology and severity of diabetic sensorimotor polyneuropathy. Eur J Neurol. 2016 Feb;23(2):354-60. doi: 10.1111/ene.12836. Epub 2015 Oct 25. PMID 26498575
- [Result] Fisse AL, Katsanos AH, Gold R, Krogias C, Pitarokoili K. Cross-sectional area reference values for peripheral nerve ultrasound in adults: A systematic review and meta-analysis-Part II: Lower extremity nerves. Eur J Neurol. 2021 Jul;28(7):2313-2318. doi: 10.1111/ene.14850. Epub 2021 May 7. PMID 33794049
- [Result] Sundaram TK. Myo-inositol catabolism in Salmonella typhimiurium: enzyme repression dependent on growth history of organism. J Gen Microbiol. 1972 Nov;73(2):209-19. doi: 10.1099/00221287-73-2-209. No abstract available. PMID 4567227
- [Result] Breiner A, Qrimli M, Ebadi H, Alabdali M, Lovblom LE, Abraham A, Albulahi H, Perkins BA, Bril V. Peripheral nerve high-resolution ultrasound in diabetes. Muscle Nerve. 2017 Feb;55(2):171-178. doi: 10.1002/mus.25223. Epub 2016 Nov 10. PMID 27312883
- [Result] Harreiter J, Roden M. [Diabetes mellitus: definition, classification, diagnosis, screening and prevention (Update 2023)]. Wien Klin Wochenschr. 2023 Jan;135(Suppl 1):7-17. doi: 10.1007/s00508-022-02122-y. Epub 2023 Apr 20. German. PMID 37101021